CLINICAL TRIAL: NCT05071612
Title: Phase 2 Randomized Double-Blind Placebo-Controlled Parallel-Arm Dose Finding Study to Compare Fixed Dose Combinations of AD109 and AD504 to Atomoxetine or Placebo in Obstructive Sleep Apnea
Brief Title: Parallel Arm Trial of AD109 and AD504 In Patients With OSA
Acronym: MARIPOSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apnimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MARIPOSA
Record Dates: First submitted 2021-09-27; First posted 2021-10-08 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: OSA - Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- AD109 Dose 1 (Experimental)
  Interventions: Drug: AD109
- AD109 Dose 2 (Experimental)
  Interventions: Drug: AD109
- AD504 Dose 1 (Experimental)
  Interventions: Drug: AD504
- AD504 Dose 2 (Experimental)
  Interventions: Drug: AD504
- Atomoxetine 1 (Active Comparator)
  Interventions: Drug: Atomoxetine Hydrochloride
- Atomoxetine 2 (Active Comparator)
  Interventions: Drug: Atomoxetine Hydrochloride
- Placebo 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AD109 — Oral administration at bedtime
  Arms: AD109 Dose 1; AD109 Dose 2
Drug: AD504 — Oral administration at bedtime
  Arms: AD504 Dose 1; AD504 Dose 2
Drug: Atomoxetine Hydrochloride — Oral administration at bedtime
  Arms: Atomoxetine 1; Atomoxetine 2
Drug: Placebo — Oral administration at bedtime
  Arms: Placebo 1; Placebo 2

SUMMARY:
This is a phase 2 randomized double-blind placebo-controlled parallel-arm dose finding study to compare fixed dose combinations of AD109 and AD504 to atomoxetine or placebo in Obstructive Sleep Apnea.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 to 65 years of age for men and 18-75 for women, inclusive, at the Screening Visit.
* Mean AHI 10 to 45 events/h, inclusive
* PGI-S: >1

Exclusion Criteria:

* Current clinically significant sleep disorder other than OSA
* Clinically significant craniofacial malformation.
* Clinically significant cardiac disease (e.g. rhythm disturbances, coronary artery disease or heart failure or hypertension requiring more than 2 medications for control).
* Participants with a history of using devices for OSA treatment, including CPAP, oral or nasal devices, or positional devices, may enroll as long as the devices have not been used for at least 2 weeks prior to first PSG and are not used during participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Change in AHI, combined AD109 dose arms vs. combined placebo arms | 28 Days
  Change in AHI (AHI, average number of events for every hour of sleep) measured by polysomnography

SECONDARY OUTCOMES:
Change in AHI, combined AD504 dose arms vs. combined placebo arms | 28 Days
  Change in AHI (AHI, average number of events for every hour of sleep) measured by polysomnography
Change in AHI, combined atomoxetine dose arms vs. combined placebo arms | 28 Days
  Change in AHI (AHI, average number of events for every hour of sleep) measured by polysomnography

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Santa Monica Clinical Trials, Los Angeles, California
  - Pacific Research Network, San Diego, California
  - SDS Clinical Trials, Inc., Santa Ana, California
  - Delta Waves, Colorado Springs, Colorado
  - Teradan Clinical Trials, Brandon, Florida
  - Research Centers of America -- Hollywood, Hollywood, Florida
  - Sleep Medicine Specialists of South Florida, Miami, Florida
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Chicago Research Center, Chicago, Illinois
  - The Center for Sleep & Wake Disorders, Chevy Chase, Maryland
  - Sleep Disorders Centers of the Mid-Atlantic (SDCMA), Glen Burnie, Maryland
  - Neurocare, Newton, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Sleep and Attention Disorders Institute, Sterling Heights, Michigan
  - Minnesota Lung Center / Minnesota Sleep Institute, Woodbury, Minnesota
  - St. Luke's Hospital Sleep Medicine, Chesterfield, Missouri
  - Clayton Sleep Institute, Maplewood, Missouri
  - Clinilabs, New York, New York
  - Coastal Carolina Health Care, P.A., New Bern, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Intrepid Research, Cincinnati, Ohio
  - Brian Abaluck, LLC, Malvern, Pennsylvania
  - Bogan Sleep Consultants LLC, Columbia, South Carolina
  - Velocity Clinical Research, Greenville, South Carolina
  - FutureSearch Trials of Neurology, Austin, Texas

REFERENCES:
- [Derived] Schweitzer PK, Taranto-Montemurro L, Ojile JM, Thein SG, Drake CL, Rosenberg R, Corser B, Abaluck B, Sangal RB, Maynard J. The Combination of Aroxybutynin and Atomoxetine in the Treatment of Obstructive Sleep Apnea (MARIPOSA): A Randomized Controlled Trial. Am J Respir Crit Care Med. 2023 Dec 15;208(12):1316-1327. doi: 10.1164/rccm.202306-1036OC. PMID 37812772